CLINICAL TRIAL: NCT05053178
Title: The Effect of Mindfulness-Based Mandala Activity on Anxiety and Spiritual Well-Being
Brief Title: The Effect of Mindfulness-Based Mandala Activity on Anxiety and Spiritual Well-Being Levels of Senior Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Çiğdem Sarı Öztürk, Dr. Cigdem Sarı Ozturk-Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2021/626
Record Dates: First submitted 2021-09-11; First posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Anxiety; Nursing Caries; ART
Keywords: art therapy; nursing student; anxiety; spirituality;
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Mindfulness-based mandala activity was applied to the intervention group via the zoom online program. Students will be divided into groups of 6-10 and mandala activities will be carried out. 3 weeks of mandala activity, breathing exercises, affirmations, etc. a therapeutic application program was created and implemented.
  Interventions: Behavioral: Mindfulness-based mandala activity
- Control group (No Intervention): For the students in the control group, the standard support program given by the school administration and course instructors will be applied for clinical problems. At the end of the study, it is planned to apply mandala activities among the students in the control group

INTERVENTIONS:
Behavioral: Mindfulness-based mandala activity — Mindfulness-based mandala activity was applied to the intervention group via the zoom online program. Students will be divided into groups of 6-10 and mandala activities will be carried out. 3 weeks of mandala activity, breathing exercises, affirmations, etc. a therapeutic application program was created and implemented
  Arms: Intervention group

SUMMARY:
This research was conducted to determine the effect of mindfulness-based mandala activity on the spiritual well-being and anxiety levels of senior nursing students in a parallel-group pretest-posttest randomized controlled study design. The required institutional permission and ethics committee approval was received. The study group of the study consisted of 170 senior nursing students (intervention group [n=84], control group [n=86]). Mindfulness-based mandala activity was applied to the intervention group via the zoom online program. Data were collected using the descriptive features form, the Spielberg Trait, and State Anxiety Inventory, the Spiritual Well-Being Scale, and the scale of the positive-negative experience. The data were stored in the SPSS 24 program.

DETAILED DESCRIPTION:
This research was conducted to determine the effect of mindfulness-based mandala activity on the spiritual well-being and anxiety levels of senior nursing students in a parallel-group pretest-posttest randomized controlled study design. The required institutional permission and ethics committee approval was received. The study group of the study consisted of 170 senior nursing students (intervention group [n=84], control group [n=86]). Mindfulness-based mandala activity was applied to the intervention group via the zoom online program. Data were collected using the descriptive features form, the Spielberg Trait, and State Anxiety Inventory, the Spiritual Well-Being Scale, and the positive-negative experiences scale. Students will be divided into groups of 6-10 and mandala activities will be carried out. 3 weeks of mandala activity, breathing exercises, affirmations, etc. a therapeutic application program was created and implemented. For the students in the control group, the standard support program given by the school administration and course instructors will be applied for clinical problems. At the end of the study, it is planned to apply mandala activities among the students in the control group. The research is based on Watson's "Human Caring" theory.

ELIGIBILITY:
Inclusion Criteria:

* Registering the theoretical and practical courses within the scope of Nursing Vocational Courses Application II,
* with internet access,
* Students who agree to participate in the study

Exclusion Criteria:

* Receiving psychiatric treatment (pharmacological and/or psychotherapy),
* with substance addiction,
* Must have participated in any meditation-based therapy program before.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Spiritual well-being scale | Change from Baseline level of Spiritual well being scale at 3 weeks (change is being assessed)
  The scale consists of 29 items and is a five-point Likert type. The lowest score of 29 points and the highest of 145 points are obtained from the scale. The higher the score indicates a higher spirituality well being.
The Spielberger State-Trait Anxiety Inventory (STAI) | Change from Baseline level of The Spielberger State-Trait Anxiety Inventory at 3 weeks (change is being assessed)
  The scale is a 40-item self-report measure of anxiety using a 4-point Likert-type scale (from 0 to 3 points) for each item. The total score obtained from the scale varies between 20 and 80. A large score indicates a high level of anxiety, and a small score indicates a low level of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sari Ozturk C, Kilicarslan Toruner E. The effect of mindfulness-based mandala activity on anxiety and spiritual well-being levels of senior nursing students: A randomized controlled study. Perspect Psychiatr Care. 2022 Oct;58(4):2897-2909. doi: 10.1111/ppc.13138. Epub 2022 Jul 3. PMID 35780483